CLINICAL TRIAL: NCT04833634
Title: Retrospective Follow-Up of the Prevision® Hip Stem in a Consecutive Case Series
Brief Title: Follow-Up of the Prevision® Hip Stem
Acronym: PRESPECT
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2008
Record Dates: First submitted 2021-04-01; First posted 2021-04-06 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Periprosthetic Fracture Around Prosthetic Joint Implant; Aseptic Loosening of Prosthetic Joint
Keywords: arthroplasty, replacement, hip; implant failure; failed primary hip arthroplasty; severe bone defects; complex bone fractures; septic loosening; poor bone remodeling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main objective of this study is to represent the treatment reality at the study site and to draw conclusions from cases of failure or suboptimal outcome. Potential risk factors for revision surgery, suboptimal outcome or radiologic sign of loosening, bone non-union or stem subsidence will be evaluated. Next to the functional outcome, stem subsidence will be used as an important indicator for a stable fixation of the revision stem.

ELIGIBILITY:
Inclusion Criteria:

* All patients implanted with a Prevision® hip stem at the study site between 2014 and 2019
* Written informed patient consent

Exclusion Criteria:

- Patients < 18 years at surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients were implanted 2-7 year before the start of the retrospective study activities.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Hip stem survival measured by Kaplan-Meier | One scheduled Follow-Up visit per patient, 2-7 years after initial implantation
  The primary endpoint of the study is hip stem survival, which is a common indicator for implant performance, which can also be used for comparison with implant registry data.

SECONDARY OUTCOMES:
Functional Outcome: Oxford Hip Score | One scheduled Follow-Up visit per patient, 2-7 years after initial implantation
  The Oxford Hip Score is a 12-item questionnaire that assesses hip function and pain. The score ranges between 12 and 60, with a lower score indicating less disability
Patient satisfaction with their endoprosthetic revision treatment | One scheduled Follow-Up visit per patient, 2-7 years after initial implantation
  The Patients are asked to grade their level of satisfaction with the outcome of the surgery at time of follow-up, with the grades: "very dissatisfied", "dissatisfied", "satisfied", "very satisfied".
  The grades may be summarized as "satisfied" vs. "dissatisfied".
Radiological evaluation (standard x-rays): Bone healing | One scheduled Follow-Up visit per patient, 2-7 years after initial implantation
  Union of the osteotomy
  o Healing of the fracture and of the greater trochanter, if applicable
Radiological evaluation (standard x-rays): osseointegration | One scheduled Follow-Up visit per patient, 2-7 years after initial implantation
  Distal and proximal radiographic bone ingrowth and Qualitative proximal remodeling
Radiological evaluation (standard x-rays): radiographic loosening | One scheduled Follow-Up visit per patient, 2-7 years after initial implantation
  Signs of radiographic loosening in the distal fixation zone
Radiological evaluation (standard x-rays): stem subsidence | One scheduled Follow-Up visit per patient, 2-7 years after initial implantation
  Stem subsidence from ap x-rays using landmarks of the femur (typically lesser trochanter) and of the prosthesis
Leg length difference | One scheduled Follow-Up visit per patient, 2-7 years after initial implantation
  Discrepancy of leg length is often considered to be a problem after total hip replacement and can adversely affect an otherwise excellent outcome and may be associated with patient dissatisfaction.
Descriptive Analysis of (Serious) adverse events | One scheduled Follow-Up visit per patient, 2-7 years after initial implantation
  (Serious) adverse events that are potentially related to the Total hip arthroplasty (THA) procedure or the THA implants will be recorded. These are events as reported by the patient, observed in the follow-up examinations or taken from the patient record

OTHER OUTCOMES:
Descriptive Analysis of Patient characteristics | One scheduled Follow-Up visit per patient, 2-7 years after initial implantation
  Age, weight, gender, date of surgery, indication for revision, comorbidities, intraoperative details

CONTACTS AND LOCATIONS:
Locations (1):
- Caritas-Krankenhaus Bad Mergentheim, Klinik für Orthopädie und Unfallchirurgie, Bad Mergentheim, Germany

REFERENCES:
- [Derived] Herold D, Kuttner A, Dreyer L, Eingartner C. Mid-term results of a cementless hip stem in femoral revision: how much diaphyseal press-fit do we need? Arch Orthop Trauma Surg. 2024 Apr;144(4):1813-1820. doi: 10.1007/s00402-023-05191-4. Epub 2024 Jan 13. PMID 38217640